CLINICAL TRIAL: NCT03495271
Title: Pilot Study of Taste Sensations in Patients With End-stage Renal Disease on Hemodialysis
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Kathleen Hill Gallant, Assistant Professor of Nutrition Science, Purdue University
Other Study IDs: 1611018504
Record Dates: First submitted 2017-11-05; First posted 2018-04-11 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Taste; Blood; Saliva
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and saliva samples collected. This is not an intervention; it is observational. Subjects will taste samples, and blood and saliva will be collected. No treatment is assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysis Patients: Inclusion Criteria:
  * Patient's undergoing hemodialysis.
  * Male and female of any race
  * 18 years/ older.
  Those with dysphagia were excluded.
  In both participant groups, before each tasting protocol commences, sterile cotton dental rolls will be placed in the participant's mouth. This will be used to collect a saliva sample and determine salivary flow.
  Tasting Protocol: The hemodialysis patients will taste each solutions twice, both before and after their dialysis session. An sensory questionnaire and an open ended comment box will be given for participants to type in other words to describe the sensations.
  In dialysis patients only, blood will be drawn pre and post dialysis for serum ion concentrations.
- Healthy Controls: Inclusion Criteria
  * No tongue, lip, or cheek piercings
  * Over 18 years of age
  * Normal taste and smell function
  * No known issues with salivation or dry mouth
  * Willing to comply with study protocol (taste samples and provide saliva)
  The above protocol will be mimicked in the healthy control group. The only difference is that instead of a pre/post dialysis tastings, the control population will have a 2-4 hour gap in between tastings in order to follow the approximate time-frame of the dialysis patients. Finally they will not be required to provide blood samples.

SUMMARY:
Individuals on dialysis due to kidney failure have very prescriptive diets. These diets help increase dialysis effectiveness and help patients control blood levels of electrolytes including potassium and phosphate, acid-base balance, blood pressure, and fluid between dialysis treatments. However, patient compliance with these diets often can be very low, and one reason for this low compliance is disguesia (abnormal taste sensations) which can make the diets unpalatable. This experiment tests the hypothesis that disguesia, and subsequent lack of adherence to a dialysis friendly diet, is a result of either vascular taste (tasting your own blood through the basolateral side of taste cells) or altered chemical composition of saliva in between dialysis appointments. However, to study these hypotheses, data are needed on the types of substances that may contribute to the disguesia. Substances for which the concentration is influenced by kidney function (in healthy people) or dialysis (in patients) are the prime candidates for the disguesia under our hypotheses. Thus, this experiment tests whether taste or flavours experienced from sodium, calcium, potassium, creatinine, urea, phosphates, glutamate, and iron may be related to altered taste experienced by patients on dialysis.

DETAILED DESCRIPTION:
A. Background:

Individuals on dialysis due to kidney failure have very prescriptive diets. These diets help increase dialysis effectiveness and help patients control blood levels of electrolytes including potassium and phosphate, acid-base balance, blood pressure, and fluid between dialysis treatments. However, patient compliance with these diets is often very low, and one reason for this low compliance is disguesia (abnormal taste sensations) which can make the diets unpalatable. The investigators hypothesize this disguesia, and subsequent lack of adherence to a dialysis friendly diet, is a result of either vascular taste (tasting one's own blood through the basolateral side of taste cells) or altered chemical composition of saliva in between dialysis appointments. However, to study these hypotheses, data are needed on the types of substances that may contribute to the disguesia. Substances for which the concentration is influenced by kidney function (in healthy people) or dialysis (in patients) are the prime candidates for the disguesia under our hypotheses.

B. Objectives:

The investigators will study how dialysis patients perceive sodium, calcium, potassium, creatinine, urea, phosphate, glutamate (umami taste), and iron solutions, and whether alterations in saliva may contribute to altered sensations from these compounds. These solutions will be used to:

1. Determine whether dialysis patients recognize the flavour of specific stimuli as similar to the disguesias experienced between dialysis treatments.
2. Determine if the intensity of the flavour from these solutions is more or less intense at the beginning of dialysis compared to the end.
3. Determine if patients' ratings for the solutions differ from healthy, control individuals.
4. Determine if saliva of patients contains different concentrations of analytes such as sodium, potassium, creatinine, urea, phosphates, iron, or glutamates from healthy controls.
5. Determine if concentrations of these analytes in saliva decrease over the course of dialysis treatment.

ELIGIBILITY:
HD subjects:

Inclusion

* Men and women
* Any race
* Age 18 years or older
* Maintenance hemodialysis patients

Exclusion

• Patients with dysphagia who are not able consume the test solutions (clear, thin liquids).

Control subjects:

Inclusion

* No tongue, lip, or cheek piercings
* Over 18 years of age
* Normal taste and smell function
* No known issues with salivation or dry mouth
* Willing to comply with study protocol (taste samples and provide saliva)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be patients (N=36) undergoing hemodialysis and healthy controls (N=36), for comparison.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Taste perception | 1 day
  Assess effect of dialysis on taste perceptions of solutions via sensory questionnaire. The scale used will be a generalized visual analog scale, which will ask participants about the intensity and hedonic quality of the sensations experienced. The scale ranges from 0 to 100 and are rated by the individuals when tasting the samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lynch KE, Lynch R, Curhan GC, Brunelli SM. Altered taste perception and nutritional status among hemodialysis patients. J Ren Nutr. 2013 Jul;23(4):288-295.e1. doi: 10.1053/j.jrn.2012.08.009. Epub 2012 Oct 6. PMID 23046735
- [Background] Seethalakshmi C, Koteeswaran D, Chiranjeevi V. Correlation of Serum and Salivary Biochemical Parameters in end Stage Renal Disease Patients Undergoing Hemodialysis in Pre and Post-Dialysis State. J Clin Diagn Res. 2014 Dec;8(12):CC12-4. doi: 10.7860/JCDR/2014/10404.5306. Epub 2014 Dec 5. PMID 25653941